CLINICAL TRIAL: NCT04888429
Title: Camrelizumab Plus Famitinib as Treatment in Patient With Advanced or Metastatic Pulmonary Sarcomatoid Carcinoma：A Multi-center, Single-arm Study
Brief Title: Camrelizumab Plus Famitinib as Treatment in Patient With Advanced or Metastatic Pulmonary Sarcomatoid Carcinoma
Acronym: CAPSTONE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qian Chu (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Qian Chu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S037
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sarcomatoid Carcinoma of Lung
Keywords: Sarcomatoid Carcinoma of Lung; Camrelizumab; Famitinib
MeSH Terms: interventions — camrelizumab; famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + Famitinib (Experimental): Patients received camrelizumab 200 mg every 3 weeks and famitinib 20 mg once per day.
  Interventions: Drug: Camrelizumab; Drug: Famitinib

INTERVENTIONS:
Drug: Camrelizumab — Patients received camrelizumab 200 mg every 3 weeks
  Other Names: SHR-1210
Drug: Famitinib — Patients received Famitinib 20 mg once per day
  Other Names: SHR-1020

SUMMARY:
This is a single arm, multi-center clinical trial. Target population is patients with Advanced or Metastatic Pulmonary Sarcomatoid Carcinoma，aiming to evaluate the efficacy and safety of the combination therapy of Camrelizumab and famitinib . Camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody, and famitinib is an orally bioavailable receptor tyrosine kinase (RTK) inhibitor.

DETAILED DESCRIPTION:
This trial enrolled patients with advanced or metastatic pulmonary sarcomatoid carcinoma. Patients will receive camrelizumab 200 mg every 3 weeks and famitinib 20 mg once per day. The primary endpoint is objective response rate (ORR) assessed by investigators per RECIST version 1.1. Key secondary endpoints were progression-free survival (PFS), overall survival (OS), duration of response, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically stage IIIB, IIIC, IV Pulmonary Sarcomatoid Carcinoma according to WHO criteria or diagnosed with non-small cell lung cancer with sarcomatoid carcinoma component (sarcomatoid component tumour cells can be spindle cells, and/or giant cells and/or heterogenous sarcomatous differentiation including rhabdomyosarcoma, chondrosarcoma, etc.) ；
* Has no prior systemic therapy; (chemotherapy and/or radiotherapy is allowed as part of neoadjuvant/adjuvant therapy. Patients who have had recurrence or metastasis for more than 6 months from the end of neoadjuvant/adjuvant treatment would be enrolled ) ；
* Patients must have at least one measurable lesion according to RECIST 1.1 ；
* ECOG score 0-1 ；
* Agree to provide tumour tissue samples for biomarker exploration (including but not limited to PD-L1 IHC or NGS testing) ；
* Life expectancy more than 3 months;
* Has adequate organ function；

Exclusion Criteria:

* Imaging (CT or MRI) showed tumor invasion of major vessels. hemoptysis ≥ 2.5 mL within 1 month before the first dose;
* Patients with EGFR-sensitive mutation (19Exondel/L858R), ALK, ROS1 gene rearrangement or fusion, BRAFV600E mutation, MET gene exon 14 skipping mutation;
* Patients with active bleeding or bleeding tendency ；
* With hypertension that cannot be reduced to the normal range after antihypertensive drug treatment (systolic blood pressure ≤ 140 mmHg/diastolic blood pressure ≤ 90 mmHg)；
* Urine protein ≥ (+ +), and 24-hour urine protein ≥ 1.0g;
* Presence of thrombotic disorder requiring anticoagulant therapy with warfarin or heparin, or requiring antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day) ；
* Has multiple factors affecting the absorption of oral drugs, such as inability to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction
* Has active central nervous system (CNS) metastases confirmed by CT or MRI
* Subjects diagnosed immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy of non-related tumor within 7 days before the first dose; allowed physiological dose of glucocorticoid (≤10 mg/day Prednisone or equivalent);
* Has active hepatitis B ;
* Has severe infections within 4 weeks of the first dose of study treatment ;
* Women who are pregnant or lactating ;
* With grade II or above myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (QTc interval ≥ 450 ms for males and QTc interval ≥ 470 ms for females). Subjects with grade III-IV cardiac insufficiency or with left ventricular ejection fraction (LVEF) less than 50% according to NYHA criteria;
* Has known history of Human Immunodeficiency Virus (HIV)；
* Has known allergy to Camrelizumab, or famitinib or any of accessories ;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | about 24 month
  Objective Response Rate using RECIST 1.1 criteria, Proportion of patients with CR and PR

SECONDARY OUTCOMES:
Progression-free Survival | about 24 month
  Time from the date of first dose to first observation of progression (RECIST1.1) or date of death (from any cause)
Overall Survival | about 24 month
  Time from the date of first dose to death from any cause
Duration of response | about 24 month
  Time from the date of the first documented response (CR or PR) to the earliest date of disease progression (RECIST 1.1), or death due to any cause.
incidence, type and severity of adverse events | From time of informed consent through treatment period and up to 30 days post last dose of study treatment (about 24 months)
  Descriptive statistics of safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Disease control rate | about 24 month
  Disease control rate using RECIST 1.1 criteria, Proportion of patients with CR, PR and SD

CONTACTS AND LOCATIONS:
Overall Officials: Qian Chu, Principal Investigator — Tongji Hospital; Lin Wu, Principal Investigator — Hunan Cancer Hospital
Locations (8):
- China (8):
  - The first Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Qian Chu, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong